CLINICAL TRIAL: NCT01313754
Title: Comparison of Skin Incision Closure Material for the Transobturator Suburethral Sling Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, David Waggonner, MD, M.D., Loma Linda University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DWSS-01
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Pain, Postoperative; Irritation (Physical); Pelvic Pain
Keywords: Skin closure; dermabond; vicryl; monocryl; Suburethral sling; Transobturator Sling; Pain; Discomfort; Skin irritation
MeSH Terms: conditions — Pain, Postoperative; Pelvic Pain; Pain | interventions — Polyglactin 910; octyl 2-cyanoacrylate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vicryl (Other): These patients will receive the standard monocryl suture on their right sided inguinal incision and then will receive the vicryl material on the left.
  Interventions: Procedure: Vicryl Suture
- Dermabond (Experimental): The patients will receive the standard monocryl suture on their right sided inguinal incision and then will receive dermabond skin glue on the left
  Interventions: Procedure: Dermabond

INTERVENTIONS:
Procedure: Vicryl Suture — Vicryl suture material will be placed on the patients left sided incision.
  Other Names: polyglactin 910
  Arms: Vicryl
Procedure: Dermabond — Dermabond skin glue will be placed on the patients left sided incision.
  Other Names: 2-octyl cyanoacrylate
  Arms: Dermabond

SUMMARY:
The purpose of this study is to compare different skin closure materials for the transobturator suburethral sling procedure. Currently the investigators are using monocryl suture material as the standard for skin closure. This material has anecdotally show to be very irritating to patients who have had this type of surgery. Our study will compare the monocryl suture material with vicryl (polyglactin 910) and dermabond (2-octyl cyanoacrylate) skin glue. The investigators believe that vicryl suture material will be superior in comfort when compared to monocryl and dermabond for this type of procedure.

ELIGIBILITY:
Inclusion Criteria:

* Those patients receiving a transobturator suburethral sling procedure.
* Adults (>= 18years).

Exclusion Criteria:

* Non-English speaking.
* Allergy to monocryl, vicryl, or dermabond.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The level of severity of patient discomfort at their incision sites. | The patients will be assessed at their second week post operative visit.

SECONDARY OUTCOMES:
Cosmesis at the incision sites | The patients will be assessed at their 2nd week post operative visit

CONTACTS AND LOCATIONS:
Overall Officials: Sam Siddighi, M.D., Principal Investigator; David B Waggonner, M.D., Study Director
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States